CLINICAL TRIAL: NCT00137137
Title: The Mini-Screw as Orthodontic Anchoring: A Clinical Trial to Study Survival, Clinical Efficiency and Experience of the Patient
Brief Title: The Mini-Screw as Orthodontic Anchoring: Survival, Clinical Efficiency and Experience of the Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/097
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Placement of the mini-screw

SUMMARY:
This is a clinical trial to evaluate the mini-screw as orthodontic anchoring. This trial will study implant survival, clinical efficiency and experience of the patient.

ELIGIBILITY:
Inclusion Criteria:

* 10-70 years of age

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Implant survival

SECONDARY OUTCOMES:
Patient opinion
Efficacy of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be